CLINICAL TRIAL: NCT00000372
Title: A Placebo Controlled Trial of Glycine Added to Clozapine in Schizophrenia
Brief Title: Glycine and D-Cycloserine in Schizophrenia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Pairing D-Cycloserine with Clozapine was found to worsen negative side effects in patients with Schizophrenia, so the study was suspended.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH057708-02 (NIH); DSIR
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
Keywords: Adult; Amino Acids; Cycloserine; Female; Glycine; Human; Male; N-Methylaspartate; Placebos; Schizophrenia; Amino Acids -- blood; Cycloserine -- *therapeutic use; Glycine -- *therapeutic use; Schizophrenia -- *drug therapy; Schizophrenia -- physiopathology
MeSH Terms: conditions — Schizophrenia | interventions — Cycloserine; Glycine; Clozapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Glycine (Experimental): The patients will undergo a 2 week single blind placebo lead in followed by an 8 week randomly assigned double blind treatment phase with 30 grams of glycine in 7 ounces of lemonade twice a day in addition to clozapine treatment.
  Interventions: Drug: Glycine; Drug: Clozapine
- Placebo (Placebo Comparator): The patients will undergo a 2 week single blind placebo lead in followed by an 8 week randomly assigned double blind treatment phase with 30 grams of placebo powder in 7 ounces of lemonade twice a day in addition to clozapine treatment.
  Interventions: Drug: Clozapine; Drug: Placebo
- D-Cycloserine (Experimental): The patients will undergo a 2 week single blind placebo lead in followed by an 8 week randomly assigned double blind treatment phase with D-cycloserine in addition to clozapine treatment.
  Interventions: Drug: D-cycloserine; Drug: Clozapine

INTERVENTIONS:
Drug: D-cycloserine
  Arms: D-Cycloserine
Drug: Glycine
  Arms: Glycine
Drug: Clozapine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects of D-cycloserine and glycine for treating negative symptoms (such as loss of interest, loss of energy, loss of warmth, and loss of humor) which occur between phases of positive symptoms (marked by hallucinations, delusions, and thought confusions) in schizophrenics.

Clozapine is currently the most effective treatment for negative symptoms of schizophrenia. Two other drugs, D-cycloserine and glycine, are being investigated as new treatments. D-cycloserine improves negative symptoms when added to some drugs, but may worsen these symptoms when given with clozapine. Glycine also improves negative symptoms and may still be able to improve these symptoms when given with clozapine. This study gives either D-cycloserine or glycine (or an inactive placebo) with clozapine to determine which is the best combination.

Patients will be assigned to 1 of 3 groups. Group 1 will receive D-cycloserine plus clozapine. Group 2 will receive glycine plus clozapine. Group 3 will receive an inactive placebo plus clozapine. Patients will receive these medications for 8 weeks. Negative symptoms of schizophrenia will be monitored through the Scale for the Assessment of Negative Symptoms, Positive symptoms will be monitored through the Positive and Negative Syndrome Scale, and additionally subjects will complete the Brief Psychiatric Rating Scale and the Global Assessment Scale.

An individual may be eligible for this study if he/she is 18 to 65 years old and has been diagnosed with schizophrenia.

DETAILED DESCRIPTION:
To determine if glycine produces improvement in negative symptoms and D-cycloserine produces worsening in symptoms compared to placebo, patients will undergo a double blind study of d-cycloserine and glycine treatment added to clozapine.

Clozapine is more effective for negative symptoms of schizophrenia than conventional neuroleptics, but the neurochemical actions contributing to this superior clinical efficacy remain unclear. Recent evidence points to a role for glutamatergic dysregulation in schizophrenia, as well as important differences between conventional agents and clozapine in effects upon glutamatergic systems. D-cycloserine, a partial agonist at the glycine modulatory site of the N-methyl-D-aspartate (NMDA) receptor, improves negative symptoms when added to conventional agents and worsens negative symptoms when added to clozapine. High-dose glycine also improves negative symptoms and has provided preliminary evidence suggesting that glycine improves negative symptoms when added to clozapine. Serum concentrations of glycine predicted response to both high-dose glycine and D-cycloserine. Both clozapine and D-cycloserine may improve negative symptoms by activation of the glycine modulatory site of the NMDA receptor complex. Because D-cycloserine is a partial agonist, it may act as an antagonist at the glycine site in the presence of clozapine, whereas the full agonist, glycine, would not be expected to worsen negative symptoms in the presence of clozapine.

This study proposes to administer a fixed-dose of D-cycloserine, glycine, or placebo added to clozapine in 45 patients with schizophrenia. Because assessments are standardized between studies, results from this study can be compared with results from a previous study of D-cycloserine added to conventional neuroleptic.

The study was ultimately suspended before participants were enrolled, due to definitive findings indicating that pairing treatment of D-cycloserine with Clozapine resulted in worsening of negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia
* Score of 27 or greater on the Scale for the Assessment of Negative Symptoms (SANS)
* Treatment with stable dose of clozapine for at least 4 weeks
* Between 18 and 65 years old

Exclusion Criteria:

* No other antipsychotic medications in oral for for at least 3 months or in depot form for 6 months
* Current major depressive episode
* Current substance abuse diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change in SANS Total Score from Baseline to Week 8 | Baseline, Week 8

SECONDARY OUTCOMES:
Change in Positive and Negative Syndrome Score from Baseline to Week 8 | Baseline, Week 8

OTHER OUTCOMES:
Change in Brief Psychotic Rating Scale from Baseline to Week 8 | Baseline, Week 8
Change in Global Assessment Scale from Baseline to Week 8 | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, MD, Principal Investigator
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Koc-Vural U, Kerimova-Kose L, Kiremitci A. Long-term clinical comparison of a resin-based composite and resin modified glass ionomer in the treatment of cervical caries lesions. Odontology. 2025 Jan;113(1):404-415. doi: 10.1007/s10266-024-00958-6. Epub 2024 Jun 5. PMID 38837034